CLINICAL TRIAL: NCT02301234
Title: Randomized, 16-Week, Multi-Phase, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Efficacy of Fulranumab as Adjunctive Therapy in Subjects With Signs and Symptoms of Osteoarthritis of the Hip or Knee
Brief Title: Study of Safety, Efficacy of Fulranumab Adjunctive Use in OA of Hip or Knee, PAI3007
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR106249; 42160443PAI3007 (Other: Janssen Research & Development, LLC); 2014-003224-40 (EudraCT Number)
Record Dates: First submitted 2014-11-21; First posted 2014-11-25 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-08

CONDITIONS: Osteoarthritis; Pain
Keywords: Osteoarthritis; Pain; Fulranumab; JNJ-42160443; Adjunctive therapy; Celecoxib; Hip; Knee; Joint replacement surgery
MeSH Terms: conditions — Osteoarthritis; Pain | interventions — fulranumab; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants will receive 4 subcutaneous (SC) injections (one injection every 4 weeks) of placebo during the double-blind treatment phase. In addition, participants may take adjunctive therapy with celecoxib 100 mg orally (by mouth) twice daily for up to 16 weeks.
  Interventions: Drug: Placebo; Drug: Celecoxib 100 mg
- Fulranumab 1 mg (Experimental): Participants will receive 4 subcutaneous (SC) injections (one injection every 4 weeks) of fulranumab 1 mg during the double-blind treatment phase. In addition, participants may take adjunctive therapy with celecoxib placebo orally twice daily for up to 16 weeks.
  Interventions: Drug: Fulranumab 1 mg; Drug: Celecoxib 100 mg Matching Placebo
- Fulranumab 3 mg (Experimental): Participants will receive 4 subcutaneous (SC) injections (one injection every 4 weeks) of fulranumab 3 mg during the double-blind treatment phase. In addition, participants may take adjunctive therapy with celecoxib placebo orally twice daily for up to 16 weeks.
  Interventions: Drug: Fulranumab 3 mg; Drug: Celecoxib 100 mg Matching Placebo

INTERVENTIONS:
Drug: Placebo — Placebo will be administered once every 4 weeks with or without adjunctive therapy for 16 weeks by subcutaneous (SC) injection (injection under the skin) into the thigh or abdomen.
  Arms: Placebo
Drug: Fulranumab 1 mg — Fulranumab will be administered once every 4 weeks with or without adjunctive therapy for up to 16 weeks by SC injection into the thigh or abdomen.
  Arms: Fulranumab 1 mg
Drug: Fulranumab 3 mg — Fulranumab will be administered once every 4 weeks with or without adjunctive therapy for up to 16 weeks by SC injection into the thigh or abdomen.
  Arms: Fulranumab 3 mg
Drug: Celecoxib 100 mg — Double-blind capsules taken twice daily for up to 16 weeks.
  Arms: Placebo
Drug: Celecoxib 100 mg Matching Placebo — Double-blind capsules taken twice daily for up to 16 weeks.
  Arms: Fulranumab 1 mg; Fulranumab 3 mg

SUMMARY:
The purpose of this study is to demonstrate the efficacy, safety, and tolerability of fulranumab as adjunctive therapy compared with placebo in participants with signs and symptoms of osteoarthritis of the hip or knee that are not adequately controlled by current pain therapy.

DETAILED DESCRIPTION:
This is a randomized (the study drug is assigned by chance), double-blind (neither physician nor participant knows the name of the assigned drug), placebo-controlled (an inactive substance is given to one group of participants while active drug is given to another group of participants to see if there is a difference in response), parallel-group (study drugs given to participants in all treatment groups during the same time period) to evaluate the efficacy (capacity of the investigational drug to produce an effect), safety, and tolerability of fulranumab administered as adjunctive therapy (in combination with other drug therapy) to participants with chronic moderate to severe pain and functional impairment from knee or hip osteoarthritis (OA) that is not adequately controlled by current pain therapy. The duration of participation in the study for an individual participant will be up to 67 weeks (includes a screening period of 3 weeks, a double-blind treatment period of 16 weeks, and a post-treatment follow-up period of up to 48 weeks). All participants will be randomly assigned in a 1:1:1 ratio to 1 of 3 treatments (placebo, fulranumab 1mg, fulranumab 3mg) and given a single injection subcutaneously (under the skin) once every 4 weeks for up to 16 weeks. In addition, participants may elect to receive adjunctive therapy (ie, double-blind supplemental oral analgesic medication or matching placebo) throughout the double-blind treatment period. Blood samples will be collected from each participant at time points during the study. Safety evaluations will include assessment of adverse events, physical examinations, laboratory tests and vital signs which will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of osteoarthritis (OA) of hip or knee based on criteria defined by the American College of Rheumatology and radiographic evidence of OA (Kellgren-Lawrence class ≥2) of the study joint
* Scheduled joint replacement or planning to undergo a joint replacement surgery for the study joint
* Unsatisfactory response (inadequate efficacy or poor tolerability) on local standard of care that includes 3 medications from at least 2 of the following classes of analgesic medications (acetaminophen/paracetamol, NSAIDs, or opioid). For participants in the USA and Canada only: Unsatisfactory response (inadequate efficacy or poor tolerability) that includes all 3 classes of analgesic medications (acetaminophen/paracetamol, NSAIDs, and opioids other than codeine or codeine combination products)
* Moderate to severe pain and functional impairment based on the NRS, WOMAC pain and physical function subscales, and PGA
* During treatment and within 24 weeks after the last injection of study drug: if female of childbearing potential, is not pregnant, breast-feeding, or planning to become pregnant, or if male, will not father a child

Exclusion Criteria:

* Increased risk of osteonecrosis (ON) or rapidly progressive osteoarthritis (RPOA)
* Unstable or progressive neurologic disorders

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2015-03-25 (Actual); Primary Completion 2016-09-19 (Actual); Study Completion 2016-09-19 (Actual)

PRIMARY OUTCOMES:
The number of participants with Adverse Events as a measure of safety and tolerability | Up to Week 52

SECONDARY OUTCOMES:
Change from baseline to the end of Week 16 in Western Ontario and McMaster University Arthritis Index (WOMAC) pain subscale score | Baseline, Week 16
  The WOMAC 3.1 is a multi-dimensional, osteoarthritis (OA) specific self-administered questionnaire using 24 questions with a 48-hour recall that are grouped into 3 subscales (pain, stiffness, and physical function) associated with hip or knee OA. Pain, stiffness, and physical function is rated on a scale of 0-10 (0 = less severe up to 10 = more severe).
Change from baseline to the end of Week 16 in Western Ontario and McMaster University Arthritis Index (WOMAC) physical function subscale score | Baseline, Week 16
  See WOMAC 3.1 described above.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (64):
- United States (32):
  - Glendale, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Anaheim, California
  - Garden Grove, California
  - Los Angeles, California
  - North Hollywood, California
  - Boulder, Colorado
  - Coral Gables, Florida
  - Miami, Florida
  - Orlando, Florida
  - Winter Park, Florida
  - Columbus, Georgia
  - Chicago, Illinois
  - Overland Park, Kansas
  - Elkridge, Maryland
  - Detroit, Michigan
  - St Louis, Missouri
  - Brooklyn, New York
  - New York, New York
  - Norman, Oklahoma
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Tullahoma, Tennessee
  - Arlington, Texas
  - Houston, Texas
  - Lampasas, Texas
  - Nassau Bay, Texas
  - Sugar Land, Texas
  - Arlington, Virginia
  - Charlottesville, Virginia
- Australia (7):
  - Camperdown
  - Hobart
  - Kippa-Ring
  - Kogarah
  - Maroochydore
  - Melbourne
  - Sherwood
- Canada (5):
  - Kamloops, British Columbia
  - Kelowna, British Columbia
  - Toronto, Ontario
  - Montreal, Quebec
  - West Vancouver
- Prague, Czechia
- Leipzig, Germany
- Szekszárd, Hungary
- Poland (6):
  - Elblag
  - Katowice
  - Krakow
  - Torun
  - Warsaw
  - Wroclaw
- South Korea (3):
  - Anyang
  - Jeju City
  - Seoul
- Spain (2):
  - A Coruña
  - Santiago de Compostela
- Sweden (2):
  - Lund
  - Malmo
- United Kingdom (4):
  - Blackpool
  - Cannock
  - Mancheter
  - Stourton

REFERENCES:
- [Derived] Kelly KM, Sanga P, Zaki N, Wang S, Haeussler J, Louie J, Thipphawong J. Safety and efficacy of fulranumab in osteoarthritis of the hip and knee: results from four early terminated phase III randomized studies. Curr Med Res Opin. 2019 Dec;35(12):2117-2127. doi: 10.1080/03007995.2019.1653068. Epub 2019 Sep 13. PMID 31387410